CLINICAL TRIAL: NCT00245284
Title: Predictor of Advanced Subclinical Atherosclerosis
Status: Completed | Type: Observational
Sponsor: PreMD (Industry)
Other Study IDs: 04K1 - PASA
Record Dates: First submitted 2005-10-26; First posted 2005-10-27 (Estimated); Last update posted 2006-06-06 (Estimated); Status verified 2006-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Evaluation of skin cholesterol for cardiovascular risk assessment in asymptomatic individuals at low, intermediate, or high risk based on Framingham Global Risk estimates. Carotid intima-media thickness (IMT), a surrogate marker for atherosclerotic burden, that independently predicts the occurrence of heart attack and stroke, will be the "gold standard" comparator.

Hypothesis: Skin cholesterol, as measured by two non-invasive tests, correlates with CAD, as measured by CIMT in this population.

DETAILED DESCRIPTION:
This study will enroll 600 asymptomatic subjects at low (<6%), intermediate (6-20% ), or high (>20%) 10-year Framingham global cardiovascular risk in approximately equal proportions.

Subjects will be enrolled from each of the three risk levels at each study site (6 total in the US). Subjects will be enrolled in a consecutive manner until there are 200 subjects from each risk level. We will track the number of subjects from each risk stratum. We will also ensure adequate representation of women (at least 33%) and African Americans (at least 25%)in the study.

We will test the subjects with 2 non-invasive skin cholesterol tests and will take a sample of blood that will be tested for serum cholesterol values and other markers of CAD. Subjects will also undego a carotid IMT scan.

The primary objective of the study is to see if skin cholesterol correlates with CAD, as measured by CIMT.

ELIGIBILITY:
Inclusion Criteria:

1. Informed written consent from the subject prior to testing.
2. Males or females 40-80 years of age

Exclusion Criteria:

1. Subjects taking cholesterol-lowering medications
2. Known hepatitis
3. Known pregnancy
4. Skin disease on either hand (e.g. eczema psoriasis, rash or broken skin)
5. Known CAD (previous myocardial infarction, coronary revascularization procedure), cerebrovascular disease (previous stroke, transient ischemic attack, or carotid revascularization procedure), or peripheral arterial disease(claudication or previous revascularization procedure)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2005-09; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: James Stein, MD, Principal Investigator — University of Wisconsin, Madison; Michael Davidson, MD, Principal Investigator — Radiant Research - Chicago; Ouyang Pamela, MD, Principal Investigator — Johns Hopkins University; Decara Jeanne, MD, Principal Investigator — University of Chicago; Mohler Emile, MD, Principal Investigator — University of Pennsylvania; Hirsch Alan, MD, Principal Investigator — University of Minnesota
Locations (6):
- United States (6):
  - Radiant Research, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - University od Pennsylvania, Philadelphia, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin